CLINICAL TRIAL: NCT02060786
Title: Point-of-Care Measurements of Platelet Inhibition After Clopidogrel Loading in Patients With Acute Coronary Syndrome: Comparison of Generic Clopidogrel Bisulfate (Plavitor®) With Original Clopidogrel Bisulfate (Plavix®)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Dong-A Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Seung-Jea Tahk, MD,PhD, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Plavitor
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Antiplatelet; clopidogrel; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- original Clopidogrel Bisulfate (Plavix®) (Active Comparator): original Clopidogrel Bisulfate (Plavix®) 600mg loading
  Interventions: Drug: original clopidogrel (Plavix® )
- generic Clopidogrel Bisulfate (Plavitor®) (Experimental): generic Clopidogrel Bisulfate (Plavitor®) 600mg loading
  Interventions: Drug: generic clopidogrel (Plavitor® )

INTERVENTIONS:
Drug: generic clopidogrel (Plavitor® )
  Arms: generic Clopidogrel Bisulfate (Plavitor®)
Drug: original clopidogrel (Plavix® )
  Arms: original Clopidogrel Bisulfate (Plavix®)

SUMMARY:
This study demonstrates the effect of generic clopidogrel bisulfate (Plavitor®) in comparison with the original clopidogrel bisulfate (Plavix®) in patients with acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unstable angina or non-ST elevation myocardial infarction
2. Patients who are planned coronary angiography
3. Age >18 years, <75 years
4. Patients who agree to the study protocol

Exclusion Criteria:

1. Recent treatment with clopidogrel or pletaal or glycoprotein IIb/IIIa Rc antagonist
2. Active bleeding (peptic ulcer, trauma or intra-cranial hemorrhage)
3. Allergy to antiplatelet agent
4. Bleeding diasthesis (blood coagulation disorders, uncontrolled severe hypertension, history of severe bleeding)
5. History of drug abuse or alcohol abuse
6. ST elevation myocardial infarction
7. Pregnancy
8. Low platelet count (< 100,000 /L) or abnormal results of PT or PTT
9. Liver disease ( bilirubin > 2 mg/dL, AST or ALT > 100 IU)
10. Renal failure ( Cr > 2.0 mg/dL)
11. Malignancy
12. Proton pump inhibitor, NSAIDs statin (except atorvastatin)

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
PRU level at 2 hours after clopidogrel loading | 2 hours after clopidogrel loading

SECONDARY OUTCOMES:
PRU level by VerifyNow P2Y12 at 4 -, 8- and 24 hours after clopidogrel loading | 4 -, 8- and 24 hours after clopidogrel loading
ARU level by VerifyNow before and 2 hours after loading | 2 hours after loading
Composite of death, myocardial infarction, target vessel revascularization | at 30 days
Stent thrombosis by Academic Research Consortium definition | at 30 days
Incidence of TIMI major bleedings | at 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, South Korea

REFERENCES:
- [Derived] Seo KW, Tahk SJ, Yang HM, Yoon MH, Shin JH, Choi SY, Lim HS, Hwang GS, Choi BJ, Park JS, Shin JS, Lee YH, Choi YW, Park SJ, Jin XJ. Point-of-care measurements of platelet inhibition after clopidogrel loading in patients with acute coronary syndrome: comparison of generic and branded clopidogrel bisulfate. Clin Ther. 2014 Nov 1;36(11):1588-94. doi: 10.1016/j.clinthera.2014.07.018. Epub 2014 Sep 15. PMID 25218311